CLINICAL TRIAL: NCT00549562
Title: A Prospective, Open-Label Study of Paliperidone ER in Adolescents and Young Adults With Autism
Brief Title: Study of Paliperidone ER in Adolescents and Young Adults With Autism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0709-24; R076477-AUT-4002
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Autism
Keywords: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paliperidone ER (Other): 8-Week Open-Label
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — Starting dose is 3 mg per day. Can be titrated up to a maximum dose of 9 mg per day.
  Other Names: Invega

SUMMARY:
This 8-week, prospective open-label study will investigate the effectiveness and tolerability of paliperidone ER in adolescents and young adults with autism. Hypothesis:Paliperidone Er will be well tolerated and efficacious for reducing aggression, self-injury, and irritability in adolescents and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between ages of 12 and 21 years
* Tanner Sage III or IV (post-pubertal)
* Diagnostic and Statistical Manual Fourth Edition Text-Revised (DSM-IV-TR) diagnosis of autism
* Outpatient
* Ability to swallow pills
* Antipsychotic medication-free for at least 2 weeks
* Score of 4 or more on the Clinical Global Impressions Severity Scale
* Score of 18 or higher on the Aberrant Behavior Checklist Irritability Scale
* Mental age of 18 months or greater based on testing
* Subjects must be in good physical health

Exclusion Criteria:

* Asperger's Disorder, Pervasive Developmental Disorder Not Otherwise Specified (PDD NOS), Rett's Disorder, childhood disintegrative disorder, schizophrenia, bipolar disorder, Fragile X Syndrome, Tuberous Sclerosis
* A significant medical condition
* An active seizure disorder
* Females who are pregnant
* Evidence of a prior adequate trial of paliperidone ER
* History of neuroleptic malignant syndrome
* Hypersensitivity to paliperidone ER

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2007-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Dunn, MD, Study Director — Indiana Univerity School of Medicine
Locations (1):
- Riley Child & Adolescent Psychiatry Clinic- Riley Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Stigler KA, Mullett JE, Erickson CA, Posey DJ, McDougle CJ. Paliperidone for irritability in adolescents and young adults with autistic disorder. Psychopharmacology (Berl). 2012 Sep;223(2):237-45. doi: 10.1007/s00213-012-2711-3. Epub 2012 May 3. PMID 22549762

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone ER: 8-Week Open-Label
  Paliperidone ER: Starting dose is 3 mg per day, with the option to increase the dose by 3 mg/day on a weekly basis for 4 weeks to a maximum dose of 12 mg per day.
Period: Overall Study
Arm/Group | Paliperidone ER
Started | 25
Completed | 23
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Years] | 15.36 [12 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 25
Clinical Global Impressions-Improvement (CGI-I) [Mean (Standard Deviation); unit: units on a scale] — The CGI Global Improvement (CGI-I) is a clinician-rate scale designed to take into account all factors to arrive at an assessment of severity and response to treatment, including parent report, parent-rated measures, teacher-rated measures, and clinician-rated measures. The CGI-I is rated from 1 to 7 (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse) at a single time-point.
  units on a scale | 4.0 (0.0)
The Aberrant Behavior Checklist [Mean (Standard Deviation); unit: units on a scale] — The Aberrant Behavior Checklist (ABC) is a 58-item measure of maladaptive behaviors and is used as a measure of drug effects. The ABC has 5 subscales:Irritability (15 items) ranging from 0 (not at all) to 45 (severe), Hyperactivity (16 items) ranging from 0 (not at all) to 48 (severe), Social Withdrawal (16 items) ranging from 0 (not at all) to 48 (severe), Stereotypy (7 items) ranging from 0 (not at all) to 21 (severe) and Inappropriate Speech (4 items) ranging from 0 (not at all) to 12 (severe). Items are rated from 0 (not at all) to 3 (severe).
  units on a scale
    ABC-Irritability | 30.3 (6.5)
    ABC-Hyperactivity | 34.7 (8.9)
    ABC-Social Withdrawal | 17.2 (12.5)
    ABC-Stereotypy | 12.5 (6.7)
    ABC-Inappropriate Speech | 7.5 (4.4)
Children's Yale-Brown Obsessive Compulsive Scale Modified for Pervasive Developmental Disorders [Mean (Standard Deviation); unit: units on a scale] — The Children's Yale-Brown Obsessive Compulsive Scale Modified for Pervasive Developmental Disorders (CY-BOCS-PDD) is semi-structured clinician rating scale designed to rate the current severity of repetitive behavior in children and adolescents with PDD. The scale consists of 5 items: Time Spent, Interference, Distress, Resistance and Control. Each item is scored from 0 (None) to 4 (Extreme). The scale yields a Total Score from 0 (least symptomatic) to 20 (most symptomatic). Higher scores indicate greater severity of repetitive behavior.
  units on a scale | 16 (3)
The Social Responsiveness Scale [Mean (Standard Deviation); unit: units on a scale] — The Social Responsiveness Scale (SRS) is a 65-item parent completed scale that assesses social awareness, social cognition, social communication, social motivation and autistic mannerisms. Each item is scored from 1 (not true) to 3 (almost always true). Interpretation in this study is based on a total score that is proportional to the level of impairment in reciprocal social behavior. Scores within 0-53 are within normal limits. Scores within 54-86 indicate mild to moderate impairment. Scores above 87 indicate severe impairment.
  units on a scale | 122.6 (18.4)
The Vineland Adaptive Behavior Scales (VABS) - Maladaptive Behavior Domain [Mean (Standard Deviation); unit: units on a scale] — The VABS Maladaptive Behavior Domain measures undesirable behaviors that may interfere with an individual's adaptive functioning. The Maladaptive Domain consists two parts. Part I contains 27 minor maladaptive items and Part II contains 9 serious maladaptive behaviors. Each item is scored from 0 (never or seldom engages in the activity) to 2(usually or habitually engages in the activity). Part 1 yields a score of 0 to 54. Part II yields a score of 0 to 18. Both parts are combined to make a Total Score of 0 to 72. High scores of maladaptive behaviors reflect more negative behavior.
  units on a scale
    VABS Maladaptive Behavior Subscale Part I | 28.9 (6.3)
    VABS Maladaptive Behavior Subscale Part II | 8.8 (6.4)
    VABS Maladaptive Behavior Subscale Total | 37.4 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: The Clinical Global Impression-Improvement(CGI-I)
Description: The CGI Global Improvement (CGI-I) is a clinician-rate scale designed to take into account all factors to arrive at an assessment of severity and response to treatment, including parent report, parent-rated measures, teacher-rated measures, and clinician-rated measures. The CGI-I is rated from 1 to 7 (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse) at a single time-point.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 25
units on a scale | 1.8 (1.3)

2. Primary Outcome: The Aberrant Behavior Checklist
Description: The Aberrant Behavior Checklist (ABC) is a 58-item measure of maladaptive behaviors and is used as a measure of drug effects. Each item is rated from 0 (not at all to 3 (severe). The ABC has 5 subscales:Irritability (15 items) ranging from 0 (not at all) to 45 (severe), Hyperactivity (16 items) ranging from 0 (not at all) to 48 (severe), Social Withdrawal (16 items) ranging from 0 (not at all) to 48 (severe), Stereotypy (7 items) ranging from 0 (not at all) to 21 (severe) and Inappropriate Speech (4 items) ranging from 0 (not at all) to 12 (severe).
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 25
units on a scale
  ABC-Irritability | 12.6 (9.1)
  ABC-Hyperactivity | 17.4 (11.5)
  ABC-Social Withdrawal | 7.6 (8.8)
  ABC-Stereotypy | 6.4 (5.1)
  ABC-Inappropriate Speech | 3.4 (3.8)

3. Secondary Outcome: The Children's Yale-Brown Obsessive Compulsive Scale Modified for Pervasive Developmental Disorders
Description: The Children's Yale-Brown Obsessive Compulsive Scale Modified for Pervasive Developmental Disorders (CY-BOCS-PDD) is semi-structured clinician rating scale designed to rate the current severity of repetitive behavior in children and adolescents with PDD. The scale consists of 5 items: Time Spent, Interference, Distress, Resistance and Control. Each item is scored from 0 (None) to 4 (Extreme). The scale yields a Total Score from 0 (least symptomatic) to 20 (most symptomatic). Higher scores indicate greater severity of repetitive behavior.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 25
units on a scale | 11.9 (4.0)

4. Secondary Outcome: The Social Responsiveness Scale
Description: The Social Responsiveness Scale (SRS) is a 65-item parent completed scale that assesses social awareness, social cognition, social communication, social motivation and autistic mannerisms. Each item is scored from 1 (not true) to 3 (almost always true). Interpretation in this study is based on a total score that is proportional to the level of impairment in reciprocal social behavior. Scores within 0-53 are within normal limits. Scores within 54-86 indicate mild to moderate impairment. Scores above 87 indicate severe impairment.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 25
units on a scale | 100.9 (20.4)

5. Secondary Outcome: The Vineland Adaptive Behavior Scales (VABS) - Maladaptive Behavior Domain
Description: The VABS Maladaptive Behavior Domain measures undesirable behaviors that may interfere with an individual's adaptive functioning. The Maladaptive Domain consists two parts. Part I contains 27 minor maladaptive items and Part II contains 9 serious maladaptive behaviors. Each item is scored from 0 (never or seldom engages in the activity) to 2(usually or habitually engages in the activity). Part 1 yields a score of 0 to 54. Part II yields a score of 0 to 18. Both parts are combined to make a Total Score of 0 to 72. High scores of maladaptive behaviors reflect more negative behavior.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 25
units on a scale
  VABS Maladaptive Behavior Subscale-Part I | 19.0 (6.9)
  VABS Maladaptive Behavior Subjscale Part II | 6.4 (3.4)
  VABS Maladaptive Behavior Subscale Total | 25.1 (8.8)

ADVERSE EVENTS:
Time Frame: Eight Weeks
Arm/Group | Paliperidone ER
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 21/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paliperidone ER (N=25)
Excessive Appetite (Gastrointestinal disorders) | 9 (9)
Weight Gain (Metabolism and nutrition disorders) | 9 (9)
Tiredness (General disorders) | 7 (7)
Rhinitis/cough (General disorders) | 8 (8)
Insomnia (Psychiatric disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Excessive saliva (General disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Enuresis (Renal and urinary disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Tic (Nervous system disorders) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1)
Dry Mouth (General disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No